CLINICAL TRIAL: NCT06437132
Title: Decoding Death and Dying in People With Dementia by Digital Thanotyping
Acronym: 5-D
Status: Recruiting | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Leiden University (Other); Harvard University (Other); Yale University (Other); Tohoku University (Other); Bergen kommune (Unknown)
Responsible Party: Principal Investigator, Bettina Husebo, Prof, MD, PhD, University of Bergen
Other Study IDs: 101088414 5-D ERC-2022-CoG
Record Dates: First submitted 2024-05-07; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Dementia
Keywords: end of life; dementia; nursing home; pain assessment and treatment; symptom assessment and treatment; mouth care
MeSH Terms: conditions — Dementia; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva and plaque collection from the mouth
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Persons with dementia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — The study is observational and will not include any specific interventions other than the regular care practice that the participants receive from their care providers. The study will use a wrist-mounted smartwatch for monitoring (Garmin VivoActive5). Previous studies show acceptability toward wearable devices among persons with dementia. Moreover, the investigator will use Somnofy, VitalThings, a radar installation mounted behind the patients bed. At the very end of life, the investigator will also apply Shimmer3 Ebio sensor measuring the patients breathing activities. Before starting the data collection, care staff will recognize any discomfort or distress potentially caused by the devices, in which case the relevant device will be immediately removed.

SUMMARY:
How can healthcare professionals recognize that a person with dementia is at the end of life? When people are dying, their physical, mental, and social abilities are gradually declining. No reliable method of predicting perceived dying currently exists although the technology is available (sensors, algorithms).

The aim of Decoding Death and Dying in Dementia by Digital thanotyping (5-D) is to provide methods and tools to diagnose and describe dying to an unprecedented level of accuracy and robustness, within a timespan larger than is possible now, focusing on the case of dying people with dementia as one of the most vulnerable and difficult to study groups. 5-D combines clinical assessment tools with wearable sensing technology to monitor a) pain and distressing symptoms, b) behavioral and psychological symptoms in dementia (BPSD), c) oral changes, and to decode "the point of no return" as the beginning of perceived dying.

To obtain this outcome in nursing home patients with dementia, the investigator will test the main hypothesis: from monitoring the evolution of thanotype components over time and their interdependencies, the prediction of the "point of no return" is possible. The objectives of 5-D are:

O1. Collect data using sensors and validated assessment scales. O2. Develop estimation methods for BPSD from sensor measurements. O3. Develop digital tools to capture the expression of pain. O4. Determine the relationship between breathing and oral symptoms. O5. Develop models for symptom interdependencies at the end of life and the "point of no return".

O6. Perform human-in-the-loop validation of developed tools, models, and algorithms.

The ground-breaking interdisciplinary novelty of 5-D endeavors to enhance the understanding of end-of-life underlying pain and symptoms in people with dementia. Advancing our theoretical knowledge to uncover how, when, and why perceived dying can be identified opens the doors for transferable research across several scientific fields

DETAILED DESCRIPTION:
Decoding death and dying in people with dementia by digital thanotyping (5-D) aims to pioneer the methodology of defining perceived dying by a data- and knowledge-driven digital representation of the end-of-life trajectory and its associated processes inferred from different measurements. The investigator proposes a novel digital thanotyping approach (Greek for thánatos) defined as the moment-by-moment in-situ quantification of the individual state of the human body. In 5-D, the investigator defines the "point of no return" as the declining state from which the person with dementia does not recover and marks the beginning of the perceived dying. In this trial the investigator describes methods and tools to define dying to an unprecedented level of accuracy and robustness, within a timespan larger than is possible now in one of the most difficult to access and vulnerable groups. Results will be transferable to other life-threatening diseases, relevant for hospitals and homecare services alike. The investigator hypothesizes that, from monitoring the evolution of clinical manifestations over time and their interdependencies, the prediction of the point of no return is possible.

5-D is a 5-year, multicenter, observation-analytic, longitudinal study aimed toward method development combining clinical data and information with systems modelling and systems identification. The investigator will recruit people with dementia (N=480) from the 10-12 Norwegian nursing homes (NH) from the Bergen Municipality, which have a cumulative capacity of >800 patients/year (out of a total of 2500 patients/year across the municipality). The recruitment pool will be extended, if necessary, to other NHs within the municipality. The investigator chooses NHs as the location for this research (instead of patient homes) because 57% of the dying population and 97% of all people with dementia in Norway die in NHs.(12) Most people in NHs present multimorbidity; among them, 52% have severe dementia (Mini-Mental-State Examination, MMSE score 0-11), 25% moderate dementia (MMSE 12-17), 16% mild dementia (18-23), and 6% no dementia (24-30).(13) Inclusion criteria: NH inhabitants >64 years, with significant cognitive impairment.(14) Exclusion criteria: people without informed/presumed consent, people already participating in other studies, people who might be distressed by sensors.

ELIGIBILITY:
Inclusion Criteria:

* Nursing home resident
* >64 years old
* People with dementia or who have a likely diagnosis of dementia
* Score of <4 on the 4 A's Test for Delirium (4AT) will be required for inclusion (no delirium)

Exclusion Criteria:

* People without dementia or cognitive impairment
* People that are considered already in a health status emergency (< 6 weeks to live)
* People that are not living in the nursing home
* People without informed/presumed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: nursing home patients with dementia
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Edmonton Symptom Assessment System (ESAS++) | Baseline and every 6.months (up to three years); When the patient is suggested to be at the end of life and is dying; ESAS will be assessed once the day.
  Symptom assessment for palliative care period and the end of life period, with added items: death rattle, dyspnea, sleep disturbances, emesis specific to end of life. Likert scale 0-10; 0 indicating no symptoms and 10 is worst symptom.
Digital biomarker estimations | Baseline and every 6.months (up to three years), continuous up to 12 weeks if a serious health event occurs]
  Digital biomarker estimations for behavioural and psychological disturbances (BPSD) e.g., apathy, agitation, pain, and sleep disturbances. Moreover, different types of breathing patterns (e.g., dyspnea, death rattle, lunge edema) Estimation of activity changes and selected BPSD resulting from the combined digital phenotype modeling; these estimations are experimental and "scores" will be based on analysis of found data after data collection period.

SECONDARY OUTCOMES:
Activities of Daily Living (ADL) - Physical Self Maintenance Scale (PSMS), Lawton and Brody, 1969. | Baseline and every 6.months (up to three years)
  Personal functional daily activities such as toileting, eating, self-care, movement/ambulation, transfers, bathing. 6 sections - scoring 1-5 on each, higher score indicates greater disability.
Neuropsychiatric Inventory - Nursing Home Version (NPI-NH) | Baseline and every 6.months (up to three years)
  Validated in Norwegian nursing homes, measuring symptoms of behavioral and psychological symptoms of dementia (BPSD) such as: apathy, agitation, depression, anxiety, sleep disturbance, and appetite/eating. Gives scores 1-4 (higher numbers being daily occurance) for amount, 1-3 for intensity and burden of care related to symptom for caregiver (1-5) for each symptom.
Mobilization - Observation - Behavioral - Intensity - Dementia Pain Scale (MOBID-2) | Baseline and every 6.months (up to three years)
  Measurement of pain specific to a dementia population; visual analog scale alongside likert scale 0-10, 0 being no pain and 10 being the worst pain, validated with persons with dementia
InterRai-Palliative Care (InterRai-PC) | Baseline and every 6.months (up to three years)
  Oral health section only/specific of the InterRai-PC, assessment of symptoms
Oral inspection | Baseline and every 4.months (up to three years)
  Biological material will be collected:
  1. for gum and mucosal tissue status, unstimulated saliva will be collected
  2. for carious lesions, collection of plaque samples will be collected from 2 teeth
  3. oral dryness will be measured using an oral moisture-checking device
  4. mucosal lesions diagnosis will be obtained from clinical pictures to determine deviation from normal healthy tissues.

OTHER OUTCOMES:
General Medical Health Rating Scale (GMHR) | Baseline
  Mortality risk measure for general wellbeing, medical comorbidity, degree of somatic illness; top 2 scores are good, bottom 2 indicate serious illness with comorbidities. Bedside measure validated in NH with people with dementia.
Chart review | Baseline
  A medication list will be compiled according to the Anatomical Therapeutic Chemical classification (ATC codes); including and of life, palliative treatment
Clinical Dementia Rating (CDR) | Baseline
  Classification of cognitive impairment, 0 no cognitive impairment, 0.5 questionable impairment, 1 mild cognitive impairment, 2 moderate cognitive impairment, 3 severe cognitive impairment.
4 A's Test for Delirium (4AT) | Baseline
  Distinction between dementia and delirium for inclusion to study, >4 indicates delirium; will be used as an exclusion criteria (participants must score <4)
Clinical Frailty Scale (CFS) | Baseline
  Mortality risk measure for general wellbeing, higher scores indicate greater disability (1-9)

CONTACTS AND LOCATIONS:
Locations (1):
- Bergen Røde Kors Sykehjem AS, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: Undecided